CLINICAL TRIAL: NCT06409130
Title: Effects of NNC0194-0499 Alone and in Combination With Semaglutide, of Semaglutide Alone, and of Cagrilintide Alone and in Combination With Semaglutide on Liver Damage and Alcohol Use in People With Alcohol-related Liver Disease
Brief Title: Effects of NNC0194-0499, Cagrilintide, and Semaglutide Alone or in Combinations on Liver Damage and Alcohol Use in People With Alcohol-related Liver Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NN9500-7730; U1111-1295-6713 (Other: World Health Organization (WHO)); 2023-508170-28 (Other: European Medical Agency (EMA))
Record Dates: First submitted 2024-05-07; First posted 2024-05-10 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Alcohol-related Liver Disease
MeSH Terms: interventions — semaglutide; cagrilintide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Sponsor staff involved in the clinical trial is masked according to company standard procedures.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (7):
- NNC0194-0499 + semaglutide (Experimental): Group A: Participants will receive subcutaneous (s.c.) injections of NNC0194-0499 in combination with semaglutide.
  Interventions: Drug: NNC0194-0499; Drug: Semaglutide
- NNC0194-0499 + semaglutide placebo (Experimental): Group A: Participants will receive subcutaneous (s.c.) injections of NNC0194-0499 in combination with semaglutide placebo.
  Interventions: Drug: NNC0194-0499; Drug: Semaglutide placebo (Group A)
- NNC0194-0499 placebo + semaglutide (Experimental): Group A: Participants will receive subcutaneous (s.c.) injections of NNC0194-0499 placebo in combination with semaglutide.
  Interventions: Drug: Semaglutide; Drug: NNC0194-0499 placebo
- NNC0194-0499 placebo + semaglutide placebo (Placebo Comparator): Group A: Participants will receive subcutaneous (s.c.) injections of NNC0194-0499 placebo in combination with semaglutide placebo.
  Interventions: Drug: NNC0194-0499 placebo; Drug: Semaglutide placebo (Group A)
- CagriSema (Experimental): Group B: Participants will receive subcutaneous (s.c.) injection of cagrilintide in combination with semaglutide.
  Interventions: Drug: Cagrilintide + semaglutide
- Cagrilintide + semaglutide placebo (Experimental): Group B: Participants will receive subcutaneous (s.c.) injection of cagrilintide in combination with semaglutide placebo.
  Interventions: Drug: Cagrilintide; Drug: Semaglutide placebo (Group B)
- Cagrilintide placebo + semaglutide placebo (Placebo Comparator): Group B: Participants will receive subcutaneous (s.c.) injection of cagrilintide placebo in combination with semaglutide placebo.
  Interventions: Drug: Cagrilintide placebo; Drug: Semaglutide placebo (Group B)

INTERVENTIONS:
Drug: NNC0194-0499 — Administered subcutaneously.
  Arms: NNC0194-0499 + semaglutide; NNC0194-0499 + semaglutide placebo
Drug: Semaglutide — Administered subcutaneously.
  Arms: NNC0194-0499 + semaglutide; NNC0194-0499 placebo + semaglutide
Drug: NNC0194-0499 placebo — Administered subcutaneously.
  Arms: NNC0194-0499 placebo + semaglutide; NNC0194-0499 placebo + semaglutide placebo
Drug: Semaglutide placebo (Group A) — Administered subcutaneously.
  Arms: NNC0194-0499 + semaglutide placebo; NNC0194-0499 placebo + semaglutide placebo
Drug: Cagrilintide + semaglutide — Administered subcutaneously.
  Arms: CagriSema
Drug: Cagrilintide — Administered subcutaneously.
  Arms: Cagrilintide + semaglutide placebo
Drug: Cagrilintide placebo — Administered subcutaneously.
  Arms: Cagrilintide placebo + semaglutide placebo
Drug: Semaglutide placebo (Group B) — Administered subcutaneously.
  Arms: Cagrilintide + semaglutide placebo; Cagrilintide placebo + semaglutide placebo

SUMMARY:
The study will look at the effects of NNC0194-0499, cagrilintide and semaglutide, on liver damage and alcohol use in participants with alcoholic liver disease. Participants will get NNC0194-0499, semaglutide, cagrilintide or ''dummy" medicine in different treatment combinations. Which treatment participants get is decided by chance. The study will last for about 39 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent obtained before any study-related activities. Study-related activities are any procedures that are carried out as part of the study, including activities to determine suitability for the study.
* Age 18 years or above, and at the legal drinking age according to local requirements at the time of signing the informed consent.
* Patient-reported history of alcohol overuse for greater than or equal to 5 years with an alcohol history of a mean of greater than or equal to 50 grams (male)/40 grams (female) pr day for the last year leading up to the time of signing informed consent.
* Enhanced Liver Fibrosis (ELF) greater than or equal to 9.0 units.

Exclusion Criteria:

* Known or suspected hypersensitivity to study intervention(s) or related products (incl. excipients).
* Previous participation (i.e., signed informed consent) in this study. If exclusion criteria 7 is met (Vibration Controlled Transient Elastography liver stiffness measurement (LSM) is greater than or equal to 25 Kilopascal (kPa)), a single rescreening is possible at the investigator's discretion.
* Documented causes of chronic liver disease other than Alcohol-related liver disease (ALD).
* Positive hepatitis B surface antigen (HBsAg), positive human immunodeficiency virus-1 (HIV-1) or HIV-2 antibody (Ab), positive hepatitis C virus (HCV) ribonucleic acid (RNA) at screening (V1) or any known presence of HCV RNA or HBsAg within 2 years of screening visit 1 (V1).
* Presence or history of ascites more than grade 1, variceal bleeding, hepatic encephalopathy, spontaneous bacterial peritonitis, or liver transplantation at screening (V1).
* Alcohol hepatitis at randomisation (as defined by National Institute on Alcohol Abuse and Alcoholism (NIAAA)).
* Vibration Controlled Transient Elastography liver stiffness measurement (LSM) greater than or equal to 25 kPa at visit 2 (V2). If participants meet this criterion, rescreening is allowed once.
* Presence or history of gastro-oesophageal varices greater than or equal to grade 2* at V2. For participants with LSM greater than or equal to 20 kPa as well as blood platelets count less than 150,000 per microliter (μL) of blood an oesophagogastroduodenoscopy performed no more than 52 weeks prior to V2 must be available at V2. *Grade 2: varices projecting by one-third of the luminal diameter that cannot be compressed with air insufflation4.
* Body mass index (BMI) less than or equal to 25 Kilogram Per Square Meter (kg/m^2).
* Female who is pregnant, breast-feeding or intends to become pregnant or is of childbearing potential and not using highly effective contraceptive method with low user-dependency.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 270 (Actual)
Dates: Start 2024-05-20 (Actual); Primary Completion 2025-11-21 (Actual); Study Completion 2026-01-16 (Actual)

PRIMARY OUTCOMES:
Change in Enhanced Liver Fibrosis (ELF) | From week 0 to week 28
  Measured as logarithm score

SECONDARY OUTCOMES:
Change in Pro-peptide of Collagen 3 (Pro-C3) | From week 0 to week 28
  Measured as ratio to baseline
Change in liver stiffness assessed by Vibration Controlled Transient Elastography (VCTE) | From week 0 to week 28
  Measured as ratio to baseline
Change in liver steatosis assessed by Controlled Attenuated Parameter (CAP) | From week 0 to week 28
  Measured as decibel milliwatts (dB/m)
Change in Alanine Aminotransferase (ALT) | From week 0 to week 28
  Measured as ratio to baseline
Change in Aspartate Aminotransferase (AST) | From week 0 to week 28
  Measured as ratio to baseline
Number of treatment emergent adverse events | From week 0 to week 35
  Measured as count of events
Change in Phosphatidylethanol (PEth) | From week -4 to week 28
  Measured as ratio to baseline
Change in alcohol amount measured by timeline followback (TLFB) | From week -4 to week 28
  Measured as grams per day
Change in total cholesterol | From week 0 to week 28
  Measured as ratio to baseline

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Transparency (dept. 2834), Study Director — Novo Nordisk A/S
Locations (102):
- United States (29):
  - The Institute for Liver Health, Chandler, Arizona
  - Arizona Liver Center, Tucson, Arizona
  - Del Sol Research Management, LLC, Tucson, Arizona
  - OM Research LLC, Lancaster, California
  - California Liver Research Institute, Pasadena, California
  - Covenant Metabolic Specialists LLC, Fort Myers, Florida
  - Miguel Rebollar PA, Hialeah, Florida
  - UF Hlth Jacksonville, Jacksonville, Florida
  - Univ of Miami/Schiff Ctr, Miami, Florida
  - Covenant Metabolic Specialists LLC, University Park, Florida
  - Rush University Med. Cntr, Chicago, Illinois
  - Kansas Medical Clinic, PA, Topeka, Kansas
  - Louisiana Research Center, LLC, Shreveport, Louisiana
  - Boston Medical Center_Cary, Boston, Massachusetts
  - Mayo Clinic Rochester, Rochester, Minnesota
  - Jubilee Clinical Research, Inc., Las Vegas, Nevada
  - DSI Research,LLC, Springboro, Ohio
  - University of Pennsylvania Hospital, Philadelphia, Pennsylvania
  - UPMC_Center for Liver Care, Pittsburgh, Pennsylvania
  - Digestive Health Research, TN, Hermitage, Tennessee
  - Texas Clinical Research Institute, Arlington, Texas
  - The Liver Institute, Dallas, Texas
  - South Texas Research Institute, Edinburg, Texas
  - Baylor St. Luke's Medical Center, Houston, Texas
  - Houston Research Institute, Houston, Texas
  - Amer. Rrsch Corp-TX Liver Inst, San Antonio, Texas
  - Pinnacle Clinical Research, San Antonio, Texas
  - Liver Specialists of Texas, Sugar Land, Texas
  - Velocity Clinical Res, Waco, Waco, Texas
- Australia (8):
  - Momentum Clinical Research Darlinghurst, Darlinghurst, New South Wales
  - Nepean Hospital, Kingswood, New South Wales
  - St George Hospital, Kogarah, New South Wales
  - Westmead Hospital, Westmead, New South Wales
  - Eastern Clinical Research Unit Box Hill, Box Hill, Victoria
  - St Vincent's Hospital (Melbourne), Fitzroy, Victoria
  - Austin Health, Heidelberg, Victoria
  - Fiona Stanley Hospital - Hepatology, Murdoch, Western Australia
- Bulgaria (6):
  - MHAT St. Ivan Rilski Gorna Oriahovitsa EOOD, Gorna Oryahovitsa
  - Acibadem City Clinic UMHAT Tokuda EAD, Gastroenterology, Sofia
  - UMHAT "Sv. Ivan Rilski", Clinic of Gastroenterology, Sofia
  - UMHAT Aleksandrovska, Sofia
  - DCC XX - Sofia EOOD, Gastroenterology, Sofia
  - Medical Center Synexus Sofia EOOD, Sofia
- Canada (5):
  - University of Calgary Liver Unit-(HMRC), Calgary, Alberta
  - GI Research Inst Foundation, Vancouver, British Columbia
  - London Health Sciences Centre- University Hospital, London, Ontario
  - TDDA Specialty Research, Vaughan, Ontario
  - Ctr de Med Metab de Lanaudiere, Terrebonne, Quebec
- Czechia (2):
  - Krajská nemocice Liberec, a.s, Liberec
  - Vseobecna Fakultni nemocnice v Praze, Prague
- Denmark (4):
  - Aalborg Universitetshospital, Aalborg
  - Herlev Hospital - Gastroenterology and Hepatology, Clinic 3, Herlev
  - Hvidovre Hospital - Gastroenheden, Hvidovre
  - Odense University Hospital - FLASH - Centre for Liver Research, Odense C
- France (3):
  - Centre Hospitalier Universitaire D'Angers-1, Angers
  - Centre Hospitalier Universitaire de Lille-Hopital Claude Huriez, Lille
  - Centre de Recherche Clinique Portes Du Sud, Vénissieux
- Germany (7):
  - Universität des Saarlandes - Innere Med. II, Homburg
  - Prof. Dr. Schiefke Ingolf, EUGASTRO GmbH, Leipzig
  - Universitätsklinikum Leipzig - Klinik und Poliklinik für Onkologie, Gastroenterologie, Hepatologie und Pneumologie, Leipzig
  - Uniklinik Schleswig-Holstein - Medizinischen Klinik I am Campus Lübeck, Lübeck
  - Universitätsmedizin der JGU Mainz - Hepatologie, Mainz
  - Universitätsklinikum Münster - Medizinische Klinik B, Münster
  - Universitätsklinikum Würzburg - Zentrum für Innere Medizin (ZIM), Würzburg
- Greece (3):
  - University Hospital of Athens ATTIKON, Athens, Attica
  - "Laiko" General Hospital of Athens, Goudi/Athens
  - 'Ippokrateio' General Hospital of Thessaloniki, Thessaloniki
- Italy (5):
  - AOU Careggi Firenze, Florence, Tuscany
  - IRCCS Ospedale Policlinico San Martino, Genova
  - Fondazione Evangelica Betania - UO Epatologia, Naples
  - Azienda Ospedaliera di Padova, Padua
  - Fondazione Policlinico Universitario Agostino Gemelli IRCS, Roma
- Japan (13):
  - Juntendo University Hospital, Gastroenterology, Bunkyo-ku, Tokyo
  - Juntendo University Hospital_Gastroenterology, Bunkyo-ku, Tokyo
  - Akaicho Clinic, Chiba-shi, Chiba
  - Ogaki Municipal Hospital_Gastroenterology and Hepatology, Gifu
  - Naka Kinen Clinic_Internal medicine, Ibaraki
  - Ishikawa Prefectural Central Hospital_Gastroenterology, Kanazawa-shi, Ishikawa
  - Kumamoto Shinto General Hospital_Liver・Gastroenterology, Kumamoto-shi, Kumamoto
  - Toranomon Hospital, Hepatology, Minato-ku, Tokyo
  - Heartlife Hospital_Liver internal medicine, Nakagamigun, Okinawa
  - Oita Cardiovascular Hospital_Gastroenterology, Oita-shi, Oita
  - JCHO Hokkaido Hospital_Digestive Disease Center, Sapporo-shi, Hokkaido
  - Saiseikai Suita Hospital, Gastroenterology, Suita-shi, Osaka
  - Nihon University Itabashi Hospital_Division of Gastro.&Hepa., Tokyo
- Netherlands (4):
  - Albert Schweitzer Ziekenhuis locatie Dordwijk, Dordrecht
  - Erasmus MC, Rotterdam
  - ETZ Elisabeth, Tilburg
  - Universitair Medisch Centrum Utrecht, Utrecht
- Poland (8):
  - Centrum Medyczne Intercor Sp. z o.o., Bydgoszcz, Kuyavian-Pomeranian Voivodeship
  - Gastromed Sp. z o.o., Torun, Kuyavian-Pomeranian Voivodeship
  - Samodzielny Publiczny Zaklad Opieki Zdrowotnej Szpital Uniwersytecki w Krakowie, Krakow, Lesser Poland Voivodeship
  - ID Clinic Arkadiusz Pisula, Myslowice, Lesser Poland Voivodeship
  - PANSTWOWY INSTYTUT MEDYCZNY MSWiA, Warsaw, Masovian Voivodeship
  - Uniwersytecki Szpital Kliniczny w Bialymstoku, Bialystok, Podlaskie Voivodeship
  - Sonomed Sp. Z O.O., Szczecin, West Pomeranian Voivodeship
  - "LANDA" Katarzyna Agata Landa, Krakow
- Spain (5):
  - Hospital Universitario Marqués de Valdecilla, Santander, Cantabria
  - Hospital Clinic i Provincial, Barcelona, Catalonia
  - Hospital Clínico Universitario de Valladolid, Valladolid, España
  - Complejo Hospitalario de Pontevedra - Hospital de Montecelo, Pontevedra, Galicia
  - Hospital Vall d'Hebron, Barcelona

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com
URL: https://novonordisk-trials.com